CLINICAL TRIAL: NCT05187260
Title: Antisense Oligonucleotide Therapy in Spinal Muscular Atrophy: An Observational Study in China
Brief Title: Antisense Oligonucleotide for Spinal Muscular Atrophy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Collaborators: Fujian Medical University Union Hospital (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wan-Jin Chen, The Director for the Department of Neurology, First Affiliated Hospital of Fujian Medical University
Other Study IDs: MRCTA,ECFAH of FMU [2021]489
Record Dates: First submitted 2021-12-25; First posted 2022-01-11 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; Antisense oligonucleotide; Neurofilament light chain
MeSH Terms: conditions — Muscular Atrophy, Spinal; Charcot-Marie-Tooth disease, Type 1F | interventions — nusinersen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5ml of CSF is collected and typically discarded as part of the typical clinical encounter when SPINRAZA® (nusinersen) is administered. This 5ml of CSF will be collected for research purposes at each dosing visit. Blood samples, including whole blood, serum, and plasma (less than 10 ml total) will be collected before intrathecal injection of SPINRAZA® (nusinersen) at each dosing visit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 5q SMA type I
  Interventions: Drug: Nusinersen
- 5q SMA type II
  Interventions: Drug: Nusinersen
- 5q SMA type III
  Interventions: Drug: Nusinersen
- Non-5q SMA
- Non-SMA subjects: Including asymptomatic carriers of SMA, relatives of SMA patients and carriers, and patients undergoing clinical standard lumbar puncture

INTERVENTIONS:
Drug: Nusinersen — SPINRAZA® (nusinersen) prescribed as part of standard of care
  Groups: 5q SMA type I; 5q SMA type II; 5q SMA type III

SUMMARY:
This is a longitudinal, multiple-center, observational study of patients genetically confirmed chromosome 5q SMA to monitor the efficacy, safety, tolerability of SPINRAZA® (nusinersen) for up to 24 months.

DETAILED DESCRIPTION:
SPINRAZA® (nusinersen) is an antisense oligonucleotide (ASO) designed to treat SMA caused by mutations in chromosome 5q that lead to SMN protein deficiency. Nusinersen, approved by the FDA for treatment of SMA in 2016, was approved by the Chinese National Medical Products Administration in 2019.

This is a prospective, longitudinal, multi-center, observational study designed to evaluate the efficacy, safety, tolerability and of nusinersen in patients genetically confirmed chromosome 5q SMA in China. Subjects with SMA I/II/III who are planning to initiate treatment with nusinersen will be enrolled in this study. All patients will be treated by their physicians according to standard clinical practice. SPINRAZA® (nusinersen) is administered as an intrathecal injection. A total of 5ml of cerebrospinal fluid (CSF) will be removed prior to administration of SPINRAZA® (nusinersen), which will be collected by the study. Neurofilament light chain (NfL) in CSF and blood will be assessed for the efficacy of nusinersen, as well as motor and pulmonary function.

There will be a total of nine visits. All the patients with 5q SMA receiving nusinersen will be visited face to face at baseline, day 14, day 28 and day 63 after treatment initiation, and then 4-month intervals through month 24/22.

ELIGIBILITY:
Inclusion Criteria:

* Patients genetically confirmed 5q SMA including types I, II and III, who are planning to initiate treatment with SPINRAZA® (nusinersen) as part of their clinical care plan.
* Non-5q SMA patients undergoing clinical standard lumbar puncture
* Non-SMA subjects including Asymptomatic carriers of SMA, relatives of SMA patients and carriers, and patients undergoing clinical standard lumbar puncture
* Participants or Parent(s)/legal guardian(s) willing and able to complete the informed consent process

Exclusion Criteria:

* Contraindication for lumbar puncture
* Inability to access intrathecal space for nusinersen injection

Ages: 1 Week to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients genetically confirmed 5q SMA including types I, II and III
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in CSF Neurofilament Light Chain levels since baseline | up to 24months
  Measured by Single-molecule Array

SECONDARY OUTCOMES:
Change in serum Neurofilament Light Chain levels since baseline | up to 24months
  Measured by Single-molecule Array

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Jin Chen, Principal Investigator — First Affiliated Hospital Fujian Medical University
Locations (3):
- China (3):
  - Department of Neurology, Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Department of Pediatrics, Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Department of Neurology, First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian